CLINICAL TRIAL: NCT02366169
Title: A Worldwide Post-Market Surveillance Registry to Assess the Medigus Ultrasonic Surgical Endostapler (MUSE™) System for the Treatment of GERD
Brief Title: Medigus Ultrasonic Surgical Endostapler (MUSE) Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medigus Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: 14-001
Record Dates: First submitted 2015-02-11; First posted 2015-02-19 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Gastroesophageal Reflux Disease (GERD)
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Medigus Ultrasonic Surgical Endostapler (MUSE) Procedure — The procedure is performed transorally under general anesthesia. The physicians staples the fundus of the stomach to the esophagus approximately 3cm superior to the Z-line in 2 or more locations. The procedural result is anatomically and functionally similar to standard anterior fundoplication (Dor-Thal operation). The staples are standard, 4.8mm titanium surgical staples. Each application of the device fires a quintuplet of staples (5) in three staggered rows. Anti-retching medications at the time of the procedure are essential.
  Other Names: Stapled anterior fundoplication

SUMMARY:
This registry is intended as an observational, post-marketing surveillance tool. The registry allows collection of baseline demographics and user experience of the commercially available MUSE system. Data collection aims to aggregate a minimum of 3 years follow-up on a large number of subjects during use outside the constraints of a prescribed clinical study.

DETAILED DESCRIPTION:
The registry evaluates the MUSE System which creates a transoral anterior fundoplication for the treatment of GERD. The system enables the operator to staple the fundus of the stomach to the esophagus approximately 3cm superior to the Z-line in 2 or more locations. The procedure is performed transorally under general anesthesia. The procedural result is anatomically and functionally similar to standard anterior fundoplication (Dor-Thal operation). The staples are standard, 4.8mm titanium surgical staples. Each application of the device fires a quintuplet of staples (5) in three staggered rows. Anti-retching medications at the time of the procedure are essential.

The study population will be primarily adults aged 18-70 years selected by the investigators based on SAGES guidelines for fundoplication and consideration of the indications and contraindications listed in the device Instructions for Use (IFU).

Follow-up data will be collected at 6 months, 1, 2 and 3 years post procedure.

ELIGIBILITY:
Inclusion Criteria:

Generally follow the guidelines for Laparoscopic Fundoplication published by SAGES (Society of American Gastrointestinal and Endoscopic Surgeons) Objective evidence of GERD

* Positive acid exposure test or endoscopic evidence of esophagitis AND
* Inadequate symptom control or
* Patient preference from surgery over medications or
* Extra-esophageal manifestations (asthma, hoarseness, cough, chest pain, aspiration)

Exclusion Criteria:

* Significant co-morbidity (for example, American Society of Anesthesiologists Grade 3 or higher)
* BMI >35 or <20
* No response to proton pump inhibitors
* Grade IV esophagitis
* Hiatal hernia >3 cm
* Irreducible hernia of any size
* Gastric outlet obstruction
* Short esophagus
* Esophageal diverticula, strictures or varices
* Esophageal motility disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The registry population will consist of adult subjects diagnosed with GERD who are deemed suitable for the procedure by the investigator given the information provided in the instructions for use.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of device and procedure related adverse events | 30 days post procedure
  Device or procedure-related adverse events and serious adverse events will be evaluated for onset, frequency and duration. The primary safety assessment time point will be within 30 days of the procedure.

SECONDARY OUTCOMES:
Procedure Durability | Up to 3 years post procedure
  Baseline and follow-up measurements of proton pump inhibitors use and GERD Health Related Quality of Life questionnaire will determine the proportion of patients with treatment success

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Kiesslich, MD, Principal Investigator — Director Klinik für Innere Medizin II; Dr. Horst Schmidt Klinik
Locations (16):
- United States (11):
  - UC Irvine Health, Orange, California
  - University of California at San Diego, San Diego, California
  - University of Florida Medical Center, Gainesville, Florida
  - The Borland Groover Clinic, Jacksonville, Florida
  - Indiana University, Indianapolis, Indiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Winthrop University Hospital, Mineola, New York
  - Lenox Hill Hospital, New York, New York
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - University of Texas Health Science Center at Houston, Houston, Texas
- Germany (3):
  - Evangelisches Krankenhaus Düsseldorf, Medizinische Klinik, Düsseldorf
  - Klinikum Ludwigsburg, Ludwigsburg
  - HSK, Dr. Horst Schmidt Kliniken GmbH, Wiesbaden
- Italy (2):
  - Ospedale San Raffaele, Milan
  - Università Cattolica del Sacro Cuore Policlinico A. Gemelli, Rome

REFERENCES:
- [Background] Zacherl J, Roy-Shapira A, Bonavina L, Bapaye A, Kiesslich R, Schoppmann SF, Kessler WR, Selzer DJ, Broderick RC, Lehman GA, Horgan S. Endoscopic anterior fundoplication with the Medigus Ultrasonic Surgical Endostapler (MUSE) for gastroesophageal reflux disease: 6-month results from a multi-center prospective trial. Surg Endosc. 2015 Jan;29(1):220-9. doi: 10.1007/s00464-014-3731-3. Epub 2014 Aug 19. PMID 25135443
- [Background] Roy-Shapira A, Bapaye A, Date S, Pujari R, Dorwat S. Trans-oral anterior fundoplication: 5-year follow-up of pilot study. Surg Endosc. 2015 Dec;29(12):3717-21. doi: 10.1007/s00464-015-4142-9. Epub 2015 Mar 18. PMID 25783833
- [Background] Kim HJ, Kwon CI, Kessler WR, Selzer DJ, McNulty G, Bapaye A, Bonavina L, Lehman GA. Long-term follow-up results of endoscopic treatment of gastroesophageal reflux disease with the MUSE endoscopic stapling device. Surg Endosc. 2016 Aug;30(8):3402-8. doi: 10.1007/s00464-015-4622-y. Epub 2015 Nov 4. PMID 26537905
- See also: Study sponsor website — http://www.medigus.com